CLINICAL TRIAL: NCT04636138
Title: Pharmacogenomic Modulators of Impaired Exercise Adaptation in Statin Users
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00145686
Record Dates: First submitted 2020-11-12; First posted 2020-11-19 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: HMG-CoA Reductase Inhibitor Toxicity
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Patients will exercise on a treadmill three times weekly at approximately 60% VO2max for 30 minutes (week one) followed by 45 minutes (week two and thereafter) for a total of 6 seeks.

SUMMARY:
3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors (statins) have beneficial effects (prevent stroke, heart attack) but also some bad ones (block some good effects of exercise). Individuals have genetic variations in proteins that metabolize/transport statins. The investigators hypothesize that these variations modulate the relationship between statin use and lack of benefit from exercise. The investigators will test this by having statin-users do supervised exercise for 6 weeks, measuring the cardiorespiratory fitness before/after and correlating this to genetic variations present in the participant.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Adults (aged 35-65 years)
* Overweight or obese (body-mass index [BMI] 25-43)
* Currently taking high-dose atorvastatin (40-80mg once daily) for primary prevention of cardiovascular disease and/or stroke
* Sedentary (<30 minutes of structured exercise weekly)
* Willing to participate in supervised exercise three times weekly
* Willing to not make intentional changes to their diet during the study period.

Exclusion Criteria:

* Tobacco smokers
* Pregnant or breastfeeding
* Use other medications that affect lipid metabolism (e.g. fibric acid, fish oil)
* Markedly functional debilitated and unable to exert 4 metabolic equivalents (METs) of energy (e.g. unable to climb a flight of stairs without stopping), or who have
* Been advised by a physician to avoid exercise due to comorbid serious cardiovascular disease
* Uncontrolled diabetes (A1c > 8)
* Uncontrolled thyroid disease
* HIV/AIDS
* Cancer
* History of myocardial infarction or stroke
* History of statin-induced myopathy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Peak oxygen consumption (VO2max) | 6 weeks
  Change pre/post intervention; compared with genomic variants

SECONDARY OUTCOMES:
Resting heart rate | 6 weeks
Resting systolic blood pressure | 6 weeks
Weight | 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J Parente, MD PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No